CLINICAL TRIAL: NCT02249845
Title: Comparing the Diagnostic Accuracy of Clinical Dehydration Scales Among Small Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Piotr Dziechciarz, MD, Medical Doctor, Medical University of Warsaw
Other Study IDs: CDS
Record Dates: First submitted 2014-09-15; First posted 2014-09-26 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Dehydration
Keywords: dehydration; children; gastroenteritis
MeSH Terms: conditions — Dehydration; Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- dehydration scales: children aged 1 - 36 months for CDS scale; 1 month - 5 years old for WHO scale and Gorelick scale

SUMMARY:
The assessment of clinical dehydration scales diagnostic accuracy (CDS scale, WHO scale, Gorelick scale) among small children.

DETAILED DESCRIPTION:
The eligible patient admitted to the hospital with acute diarrhea, after given written consent for participation in the study by the child's parents, will be clinically assessed. Dehydration syndromes noted by physician will be recorded in special form (in attachment). Than, the child will be weighted on a standard scale.

The next body mass evaluation will take place, when patient's clinical condition will by classified as good by the attending physician and the child will be at least 24 hours after finishing intravenous or probe rehydration therapy.

ELIGIBILITY:
Inclusion Criteria:

* age: 1 - 36 months for CDS scale; 1 month - 5 years old for WHO scale and Gorelick scale
* hospitalisation caused by acute diarrhea (acute diarrhea -increase in the frequency of evacuations ≥ 3 in 24 hours; with or without fever or vomiting)
* duration of symptoms under 5 days
* parents' written consent for child's participation in the study

Exclusion Criteria:

* Dehydration caused by other mechanisms than acute diarrhea, for example dehydration caused by:

  * acidosis
  * kidney failure
  * heart failure
  * chronic liver disease
  * respiratory failure
  * condition after surgery

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Small children with acute diarrhoea admitted to the pediatric ward.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
CDS scale evaluation | all necessary data will be collected till patient's discharge day (ca. 5 days after admition to the hospital)
  sensitivity, specificity, positive and negative likelihood ratios for CDS scale for dehydration <3%, 3-6%, >6%
WHO scale evaluation | all necessary data will be collected till patient's discharge day (ca. 5 days after admition to the hospital)
  sensitivity, specificity, positive and negative likelihood ratios for WHO scale for dehydration <5%, 5-10%, >10%
Gorelick scale evaluation | when all data will be collectedall necessary data will be collected till patient's discharge day (ca. 5 days after admition to the hospital)
  sensitivity, specificity, positive and negative likelihood ratios for Gorelick scale for dehydration ≥5%, ≥10%

CONTACTS AND LOCATIONS:
Overall Officials: Anna Falszewska, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Pediatrics, Medical University of Warsaw, Warsaw, Poland